CLINICAL TRIAL: NCT07388667
Title: A Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MK-4082 in Healthy Overweight/Obese Participants
Brief Title: A Clinical Study of MK-4082 in Healthy Overweight Participants (MK-4082-002)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: 4082-002; MK-4082-002 (Other: MSD)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Panel A: Dose Escalation to Dosage 1 (Experimental): Participants receive escalating doses of oral MK-4082 once daily (QD) or a dose-matched placebo to reach maintenance dose 1.
  Interventions: Drug: MK-4082; Drug: Placebo
- Panel B: Dose Escalation to Dosage 2 (Experimental): Participants receive escalating doses of oral MK-4082 QD or a dose-matched placebo to reach maintenance dose 2.
  Interventions: Drug: MK-4082; Drug: Placebo
- Panel C: Dose Escalation to Dosage 3 (Experimental): Participants receive escalating doses of oral MK-4082 once daily (QD) or a dose-matched placebo to reach maintenance dose 3.
  Interventions: Drug: MK-4082; Drug: Placebo
- Panel D: Dose Escalation to Dosage 4 (Experimental): Participants receive escalating doses of oral MK-4082 once daily (QD) or a dose-matched placebo to reach maintenance dose 4.
  Interventions: Drug: MK-4082; Drug: Placebo
- Panel E: Dose Escalation to Dosage 5 (Experimental): Participants receive escalating doses of oral MK-4082 once daily (QD) or a dose-matched placebo to reach maintenance dose 5.
  Interventions: Drug: MK-4082; Drug: Placebo

INTERVENTIONS:
Drug: MK-4082 — Oral Tablet
Drug: Placebo — Oral Tablet

SUMMARY:
Researchers are looking for new weight loss medicines for people with higher body weight. The study medicine, MK-4082, is different from similar weight loss medicines because people take it as a pill instead of an injection. Before giving a study medicine to people with a health condition, researchers first do studies to find a safe dose level (amount) of the study medicine that can be used in future studies.

The goals of this study are to learn about:

* The safety of MK-4082 and if people tolerate it
* What happens to different MK-4082 dose levels in a person's body over time

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is in good health
* Has body mass index (BMI) between 25 and 40 kg/m^2, inclusive. Participants must weigh at least 60 kg

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* has a history of previous surgical treatment for obesity (bariatric surgery, gastric banding, etc.) or any other gastrointestinal (GI) surgery that may induce malabsorption, history of bowel resection >20 cm, any malabsorption disorder, severe gastroparesis, or any GI procedure for weight loss (including LAP-BAND®), as well as clinically significant GI disorders (eg, peptic ulcers, severe gastroesophageal reflux disease)
* has an individual or family history of medullary thyroid carcinoma or multiple endocrine neoplasia 2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 98 Days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 84 Days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Curve from Time 0 to 24 hours (AUC0-24) of MK-4082 | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24hr of MK-4082.
Time to Maximum Plasma Concentration (Tmax) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the Tmax of MK-4082.
Maximum Plasma Concentration (Cmax) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the Cmax of MK-4082.
Plasma Concentration at 24 Hours (C24) of MK-4082 | At designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the C24 of MK-4082.
Area Under the Curve from Time 0 to Infinity (AUC0-Inf) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the AUC0-Inf of MK-4082.
Area Under the Curve from Time 0 to Last (AUC0-Last) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the AUC0-last of MK-4082.
Apparent Clearance (CL/F) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the CL/F of MK-4082.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the Vz/F of MK-4082.
Apparent Terminal Half-life (t1/2) of MK-4082 | Predose and at designated timepoints up to 84 Days postdose
  Blood samples will be collected to determine the t1/2of MK-4082.
Change from Baseline in Body Weight | Baseline and up to approximately 84 Days
  Change from baseline in body weight will be reported.
Change from Baseline in Body Mass Index (BMI) | Baseline and up to approximately 84 Days
  Change from baseline in body mass index (BMI) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com